CLINICAL TRIAL: NCT04767308
Title: A Single-center, Single-arm Exploratory Clinical Trial to Evaluate the Safety and Efficacy of Fully Human Anti-CD5 Chimeric Antigen Receptor T Cells (CT125A Cells) for the Treatment of Relapsed/Refractory CD5+ Hematopoietic Malignancies
Brief Title: Safety and Efficacy of CT125A Cells for Treatment of Relapsed/Refractory CD5+ Hematopoietic Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Shanghai IASO Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jianfeng Zhou, Principal Investigator, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT125ACI001
Record Dates: First submitted 2021-02-09; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: CD5+ Relapsed/Refractory Hematopoietic Malignancies; Chronic Lymphocytic Leukemia (CLL); Mantle Cell Lymphoma (MCL); Diffuse Large B-cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Peripheral T-cell Lymphomas (PTCL)
Keywords: Adoptive T Cell Therapy; Chimeric antigen receptor; CD5 / Lymphocyte antigen T1/Leu-1; CD5+ hematopoietic malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, T-Cell, Peripheral | interventions — CF regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): The tolerability and safety of CT125A cells will be assessed according to the "3+3" dose escalation design. There will be three dose levels, 1×10^6, 2×10^6, and 3×10^6, CAR+T cells/kg. For each level, 1-3 subjects will be enrolled. If no dose limited toxicity (DLT) occurs, next level will be assessed for DLT. If DLT occurs in one subject, 3 more subjects will be enrolled in this cohort for the evaluation of DLT. If DLT occurs in ≤ 1/6 subjects, next level will be assessed for DLT. If DLT occurs in ≥ 2 subjects, no more subjects will be enrolled in this cohort and dose escalation will be canceled. For each cohort, following subjects can only receive CT125A infusion at least 14 days after the first subject received CT125A infusion. If DLT occurs in 2 subjects at Dose Level 1, whether to explore a lower dose will be determined by the investigator. After dose escalation phase is completed, the dose for extension phase will be determined based on safety and PK data.
  Interventions: Biological: CT125A cells; Drug: Cyclophosphamide, fludarabine

INTERVENTIONS:
Biological: CT125A cells — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to manufacture CT125A cells, during which cyclophosphamide and fludarabine will be administered for the purpose of lymphocytes depletion. After lymphodepletion, subjects will receive one dose treatment with CT125A cells by intravenous (IV) infusion. The initial dose of 1×10^6 CAR+ T cells/kg will be infused on day 0.
Drug: Cyclophosphamide, fludarabine — Subjects will be given IV infusion of cyclophosphamide 500 mg/m2/day and fludarabine 30 mg/m2/day on days -4, -3 and -2

SUMMARY:
Current treatments for relapsed/refractory hematopoietic malignancies such as B-cell lymphomas (BCLs) and peripheral T-cell lymphomas (PTCLs) are far from satisfactory. CD5 is widely expressed in multiple subtypes of BCLs and PTCLs but rarely found in normal tissues except certain types of lymphocytes. Chimeric antigen receptor (CAR) T cells against CD5 offer another potential therapeutic option for patients with relapsed/refractory CD5 positive hematopoietic malignancies. In the current study, the safety and efficacy of a novel CAR T cell therapy, termed CT125A cells, are evaluated in patients with relapsed/refractory CD5+ hematopoietic malignancies. The endogenous CD5 in CT125A cells is knocked out via CRISPR/Cas9 genome editing technology to prevent fratricide during CAR T cells manufacturing.

ELIGIBILITY:
Inclusion Criteria:

1.Subjects with CD5 positive B-cell lymphomas must meet the diagnostic criteria from National Comprehensive Cancer Network (NCCN) guidelines for B-Cell Lymphomas (2020.V1) and have CD5 expression on lymphoma cells (results within 60 days before informed consent signing are acceptable if current clinical condition is not suitable for sampling, and the investigator will judge whether the test results from other hospitals are acceptable and whether they can be enrolled); according to Lugano 2014 criteria, patients with B-cell lymphomas have at least one measurable lesion with the longest diameter ≥ 1.5 cm or bone marrow involvement detected by flow cytometry .

Including:

1. Chronic lymphocytic leukemia/small lymphocytic lymphoma: any BTK inhibitor have been given for at least 6 months and the treatment has failed (SD or PD).
2. Mantle cell lymphoma (MCL): patients with MCL must have relapsed/refractory diseases after receiving at least one treatment regimen. Previous treatment must include chemotherapy with anthracyclines or bendamustine, anti-CD20 monoclonal antibody, and any BTK Inhibitor therapy.
3. Diffuse large B-cell lymphoma: patients with diffuse large B-cell lymphoma who have failed or relapsed after at least two lines of therapy (a standard chemotherapy and a rescue chemotherapy); and meet one of the following conditions: a. unable to receive autologous hematopoietic stem cell transplantation (autoHSCT); b. refuse to receive autoHSCT; c. relapse after autoHSCT.

2.Subjects with CD5 positive peripheral T-cell lymphomas (PTCLs) are diagnosed according to criteria from World Health Organization classification for tumors of the hematopoietic and lymphoid tissues (2016 Edition) and have CD5 expression on lymphoma cells (results within 60 days before informed consent signing are acceptable if current clinical condition is not suitable for sampling, and the investigator will judge whether the test results from other hospitals are acceptable and whether they can be enrolled); according to Lugano 2014 criteria, patients with T-cell lymphomas must have at least one measurable lesion with the longest diameter ≥ 1.5 cm and no bone marrow involvement confirmed by flow cytometry and gene rearrangement (TCR/IGH) tests (and PET-CT results, if any, that must indicate no increased bone marrow metabolism); patients must fail or relapse after at least one line of therapy; including but not limited to the following PTCLs:

1. Peripheral T cell lymphoma - not otherwise specified (PTCL-NOS)
2. Angioimmunoblastic lymphoma
3. ALK negative anaplastic large cell lymphoma
4. Extranodal NK/T cell lymphoma
5. Enteropathy-associated T-cell lymphoma
6. Large granular T lymphocyte leukemia
7. Adult T cell leukemia

3.Age ≥18 and ≤70 years old, regardless of gender.

4.Expected life expectancy ≥12 weeks.

5.Serum total bilirubin ≤ 37.2 μmol/L (Gilbert syndrome patients ≤ 3.0 ULN, direct bilirubin ≤ 1.5 ULN), estimated glomerular filtration rate eGFR (CKD-EPI) ≥ 30 ml/min/1.73m2, alanine aminotransferase and aspartate aminotransferase less than 2.5 times the upper limit of normal range.

6.ECOG score 0-1 points.

7.Echocardiography suggests left ventricular ejection fraction (LVEF) ≥50%; blood oxygen saturation >91%.

8.After signing the informed consent form, subjects and their partners must be willing to use effective and reliable method of contraception, devices or medicines, within one year after CAR T cell infusion (excluding contraception safety periods). A negative pregnancy test must be obtained for female subjects.

Subjects must provide written informed consent before the study begin.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded:

1. History of allergies to any of the ingredients in cell products.
2. Patients with acute GVHD judged to be grade II-Ⅳ by Glucksberg criteria or grade B-D by IBMTR index; acute or chronic GVHD patients who need systemic treatment within four weeks before enrollment.
3. Injected with live vaccines within 4 weeks before enrollment.
4. Central nervous system diseases not associated with lymphoma CNS invasion (such as cerebral aneurysm, epilepsy, stroke, senile dementia, psychosis, etc.). Lymphoma CNS invasion or digestive tract invasion is not considered as an exclusion criterion, but whether to be enrolled in the group is determined by the investigator.
5. Severe active infection (except simple urinary tract infection and bacterial pharyngitis), or currently receiving intravenous antibiotic treatment. However, preventive antibiotics, antiviral and antifungal infection treatments are permitted.
6. Hepatitis B surface antigen (HBsAg) positive or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA > 100 IU/mL.
7. Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive.
8. Subjects with other acquired and congenital immunodeficiency diseases, including but not limited to human immunodeficiency virus (HIV) antibody positive; subjects with cytomegalovirus (CMV) DNA > 400 copy/mL; subjects with syphilis test positive.
9. Cardiac insufficiency of grade III or IV according to the New York Heart Association (NYHA) cardiac function classification criteria.
10. History of other primary cancers, except for the following conditions:

1)Non-melanoma skin cancer with complete resection, such as basal cell carcinoma; 2)Cured carcinoma in situ such as cervical cancer, bladder cancer or breast cancer; 3)No recurrence of other primary cancers has been found for more than 5 years after treatment.

11.History of solid organ transplantation.

12.Subjects with previous autoimmune diseases (mainly abnormality of cellular immunity), immunodeficiency or subjects requiring immunosuppressive therapy.

13.Received other interventional clinical trial treatment within 3 months before signing ICF.

14.Pregnant or lactating women.

15.Suffer from mental illness or disturbance of consciousness or central nervous system disease.

16.The toxicity of previous treatment has not been relieved to baseline or ≤2 (NCI-CTCAE v5.0, except for hair loss).

17.Drug use:

1. Steroid drugs: therapeutic dose of steroids used within 72 hours before CAR-T cell infusion, but physiological doses of steroid supplementation are allowed (<12mg/m2/day of hydrocortisone or its equivalent dose);
2. Systemic anti-tumor therapy is not ended at least 2 weeks or 5 drug half-lives before apheresis (except for BTK inhibitors in CLL); interval between apheresis and immune checkpoint inhibitor treatment is less than 3 drug half-lives.

18.Active lung infection.

19.Contraindications for peripheral blood apheresis.

20. Subjects considered unsuitable for enrollment by the investigator for other reasons after careful consideration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and types of dose limited toxicities (DLTs) following infusion of CT125A chimeric antigen receptor (CAR) T cells | 28 days after CAR T cell infusion
  Incidence and types of dose limited toxicities (DLTs) after administration of CT125A cells in patients with relapsed/refractory CD5+ hematopoietic malignancies will be recorded at 3 dose levels to investigate the maximum tolerated dose of CT125A. DLT is defined as the following adverse events that occur during the first 28 days after CT125A infusion and are definitely or probably related to CT125A cells: 1) Cytokine release syndrome equal or greater than grade 4 lasting longer than 3 days graded by ASTCT 2019 consensus; 2) Grade 4 immune effector cell-associated neurotoxicity syndrome graded by ASTCT 2019 consensus; 3) Grade 4 hematological toxicity lasting longer than 28 days except for T cell aplasia; 4) Non-hematological toxicity equal or greater than grade 3 lasting longer than 7 days or Grade 4 non-hematological toxicity lasting longer than 3 days.
Incidence and severity of adverse events (AEs) following infusion of CT125A chimeric antigen receptor (CAR) T cells | 2 years after CAR T cell infusion
  Incidence of adverse events (AEs) after administration of each dose of CT125A cells in patients with relapsed/refractory CD5+ hematopoietic malignancies will be recorded and the severity of AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 except that cytokine release syndrome and immune effector cell-associated neurotoxicity syndrome will be graded according to the consensus by ASTCT in 2019. AE is defined as any untoward medical occurrence in a patient after CAR T cell infusion and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Overall response rate (ORR) at 4th week and 12th week | 12 weeks after CAR T cell infusion
  At 4 weeks and 12 weeks after CT125A infusion, the response rate of subjects that are evaluated as complete response (CR) and partial response (PR) according to Lugano 2014 criteria will be measured
Time to first response after CT125A cells infusion | 2 years after CAR T cell infusion
  The number of days elapsed between the time when subjects receive CT125A infusion and the time when the response is first evaluated as partial response (PR) or complete response (CR) will be measured
Time to complete response (CR) after CT125A infusion | 2 years after CAR T cell infusion
  The number of days elapsed between the time when subjects receive CT125A infusion and the time when the response is first evaluated as complete response (CR) will be measured

OTHER OUTCOMES:
Best overall response (BOR) 3 months after CT125A cells infusion | 3 months after CAR T cell infusion
  Within 3 months after CT125A infusion, the percentage of subjects whose best responses are evaluated as partial response (PR) or complete response (CR) will be measured
Duration of response (DOR) | 2 years after CAR T cell infusion
  The number of days between the time when the response is first evaluated as CR or PR after CT125A infusion and the time when the subject is first evaluated to have progressive disease (PD) or dies for any reason
Progression free survival (PFS) | 2 years after CAR T cell infusion
  The number of days between the time when subjects receive CT125A infusion and the time when the subject is first evaluated to have progressive disease (PD) or dies for any reason
Overall survival (OS) | 2 years after CAR T cell infusion
  The number of days between the time when subjects receive CT125A infusion and the time when subjects die for any reason
Quantification of vector copy number (VCN) in peripheral blood following CT125A infusion by ddPCR | 2 years after CAR T cell infusion
  The vector copy number (VCN) of CAR transgene measured as copies per microgram of genomic DNA in peripheral blood will be determined by droplet digital polymerase chain reaction (ddPCR) analysis before CT125A infusion; on day 0, 1, 4, 7, 11, 14, 21, and 28; week 8, 12, 24, and 36; and every 3 month 9 months after CT125A infusion. The kinetics of VCN will be plotted to assess the expansion and persistence of CAR T cells.
Assessment of CAR T cells expansion in peripheral blood or bone marrow following CT125A infusion by flow cytometry | 2 years after CAR T cell infusion
  The absolute number of CAR T cells per milli-liter of peripheral blood will be determined by flow cytometry analysis and absolute lymphocyte count test before CT125A infusion; on day 0, 1, 4, 7, 11, 14, 21, and 28; week 8, 12, 24, and 36; and every 3 month 9 months after CT125A infusion. The kinetics of CT125A cells will be plotted to assess the expansion and persistence of CAR T cells.
Evaluation of the dynamic changes of lymphocytes before and after CT125A infusion by flow cytometry | 2 years after CAR T cell infusion
  The subsets of lymphocytes and the number of CD5 positive cells in peripheral blood will be determined by flow cytometry analysis before CT125A infusion; on day 0, 1, 4, 7, 11, 14, 21, and 28; week 8, 12, 24, and 36; and every 3 month 9 months after CT125A infusion. The relative abundance (percentage of total leukocytes) or absolute number (number per milli-liter) of lymphocyte subsets will be measured by flow cytometry analysis and absolute lymphocyte count test.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhou, PhD, MD, Principal Investigator — Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data that underlie the results published will be shared in the publication. Data will be available upon request and after the approval of data request proposal.

REFERENCES:
- [Derived] Cheng J, Zhu L, Wu J, Zeng Y, Mao X, Ding S, Wang J, Xiao Y, Zhou X, Mu W, Zhu X. Efficacy and safety of autologous CD5-KO anti-CD5 CAR-T cells in relapsed/refractory CD5+ hematological malignancies. Cell Rep Med. 2026 Feb 2:102584. doi: 10.1016/j.xcrm.2026.102584. Online ahead of print. PMID 41633358
- [Derived] Mu W, Zhang M, Hu G, Han Y, Mao X, Chen C, Shen K, Dai Z, Zhu X, Zhou X, Huang L, Ao Q, Xiao M. Case report: Differential diagnosis of highly amplified anti-CD5 CAR T cells and relapsed lymphoma cells in a patient with refractory ALK positive anaplastic large cell lymphoma. Front Immunol. 2023 Dec 8;14:1280007. doi: 10.3389/fimmu.2023.1280007. eCollection 2023. PMID 38143760